CLINICAL TRIAL: NCT06114940
Title: PLUTO: A Prospective Phase II Study of Perioperative TORIPALIMAB Plus LENVATINIB in Patients With Renal Cell Carcinoma Undergoing Nephrectomy
Brief Title: Perioperative TORIPALIMAB Plus LENVATINIB in Patients With Renal Cell Carcinoma Undergoing Nephrectomy (PLUTO)
Acronym: PLUTO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Le Qu, Associate chief urologist, Jinling Hospital, China
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2025DZKY-005-02
Record Dates: First submitted 2023-09-03; First posted 2023-11-02 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Renal Cell Carcinoma (RCC)
Keywords: ccRCC; Perioperative therapy; Immunotherapy; Tyrosine Kinase Inhibitors; nephrectomy
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — toripalimab; spartalizumab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Toripalimab + Lenvatinib followed by nephrectomy (Experimental): After 4-5 cycles of preoperative therapy, patients will undergo nephrectomy within 4 weeks. Patients with WHO/ISUP grading 4 RCC in cohort 1, and all patients of cohort 2 and 3 will receive postoperative dosing within 4 weeks for at most 17 doses. Subsequent follow-up will then be completed to assess adverse events and long-term outcomes.
  Cohort 1: Localized RCC (cT1b-T2bN0M0). Nephrectomy following preoperative therapy. For patients with WHO/ISUP grading 4 RCC in the resected tumor, postoperative dosing of Toripalimab beginning within 4 weeks after surgery for at most 17 doses.
  Cohort 2: Locally advanced RCC (cT3-4N0M0 or cTanyN1M0). Nephrectomy following preoperative therapy. Postoperative dosing of Toripalimab beginning within 4 weeks after surgery for at most 17 doses.
  Cohort 3: Metastatic RCC (cTanyNanyM1). Cytoreductive nephrectomy following preoperative therapy. Postoperative dosing of Toripalimab plus Lenvatinib beginning within 4 weeks after surgery for at most 17 doses.
  Interventions: Drug: Toripalimab; Drug: Lenvatinib

INTERVENTIONS:
Drug: Toripalimab — Preoperative: Toripalimab 240mg, IV on day 1 in a 3-week cycle. Preoperative Toripalimab contains 4-5 cycles.
  Postoperative: Toripalimab 240mg, IV on day 1 of a 3-week cycle. Postoperative Toripalimab following surgery within 4 weeks for patients mentioned above in cohort 1, 2 and 3.
  Other Names: anti-PD-1 monoclonal antibody
Drug: Lenvatinib — Preoperative: Lenvatinib 20 mg orally, QD in a 3-week cycle. Preoperative Lenvatinib contains 4-5 cycles.
  Postoperative: Lenvatinib 20 mg orally, QD in a 3-week cycle. Postoperative Lenvatinib following surgery within 4 weeks for patients in cohort 3.
  Adjustment of dose: For patients with intolerable adverse reactions (CTCAE v5.0 grade 3 or grater), the dose could be reduced to 12mg for those who were suitable to continue taking the drug after systematic evaluation by the investigator. Patients who are assessed as intolerable and not suitable for continued medication will discontinue and undergo nephrectomy within 4 weeks.
  Other Names: Lenvatinib mesylate (USAN); E7080; ER-203492-00; Multi-Kinase Inhibitor E7080

SUMMARY:
The PLUTO-trial is a single-center, open-label, phase II trial investigating Toripalimab plus Lenvatinib in patients with multi-stage clear-cell renal cell carcinoma. In this trial, patients will be enrolled in one of three cohorts according to the stage of their clear-cell renal-cell carcinoma: localized, locally advanced and metastatic RCC. Patients in all cohorts will receive four to five cycles of preoperative Toripalimab (240mg Q3W IV) plus Lenvatinib (20mg QD PO) and will undergo nephrectomy within four weeks after the last cycle. Patients in cohort 1 who are considered to be at high risk according to pathology results of surgery specimen, and all the patients in cohort 2 are supposed to receive postoperative doses of Toripalimab (240mg Q3W IV) for at most 17 doses. Patients in cohort 3 are supposed to continue Toripalimab plus Lenvatinib after surgery.

The primary clinical endpoint of the study is immune-related pathological response to tumorigenesis, defined as the extent of tumor cell reduction in the tumor bed. Simon's two-stage design is used in this study. An initial cohort of 12 patients per cohort will be recruited, followed by an interim analysis. Recruitment to each cohort will be closed if a qualifying immune-related pathological response is not observed in any patient at an interim analysis. If qualifying immune-related pathological response is observed in at least one patient, additional 9 patients will be recruited in the cohort to 21 patients. Considering potential 10% dropout rate in the trial, an anticipation of 69 patients will be recruited for this study.

ELIGIBILITY:
Inclusion Criteria:

* Have fully understood and voluntarily signed the informed consent Form (ICF);
* Age: 18-80 years old (at the time of signing the informed consent); Both male and female; ECOG PS score: 0-1;
* RCC with clear cell component confirmed by histology or cytopathology, including locally advanced RCC with clear cell component;
* ECOG 0-1 points
* T1b-T2bN0M0, T3a-4N0M0, TanyN1M0 or M1RCC diagnosed by imaging at initial diagnosis:

  1. Cohort 1: T1b-T2bN0M0 RCC;
  2. Cohort 2: T3a-4N0M0 or TanyN1M0 RCC;
  3. Cohort 3: M1 RCC undergoing cytoreductive nephrectomy.
* Radical nephrectomy or partial nephrectomy or renal tumor enucleation was decided after the clinician made the treatment plan and communicated with the patient;
* Willingness and ability to comply with planned visits, therapeutic laboratory testing, and other procedures.

Exclusion Criteria:

* Signs of tumor metastasis involving the central nervous system;
* History of malignant tumors other than the study disease within the previous 5 years, with the exception of malignant tumors that can be expected to be cured with treatment (including but not limited to adequately treated thyroid cancer, carcinoma in situ of the cervix, basal or squamous cell skin cancer, or ductal carcinoma in situ of the breast treated with radical surgery);
* Prior to participating in the study, patients had received other systemic treatment drugs, including targeted drugs, immunotherapy drugs and their combination regimens, or local anti-tumor therapy, or received investigational drugs or device therapy;
* Underwent major surgery (judged by the investigator) within 4 weeks before the first trial dose, were recovering, or were unable to undergo baseline puncture;
* History of severe drug allergy, including but not limited to antibody drugs;
* patients with contraindications to immunotherapy restart, including but not limited to:

  1. Grade 2-4 immune myocarditis;
  2. Severe grade 4 proteinuria;
  3. Severe or life-threatening grade 4 immune hepatitis;
  4. Severe grade 3-4 immune pneumonitis;
  5. Severe inflammatory arthritis that significantly affects daily life or quality of life;
  6. Severe neurological toxicity:
  7. Myasthenia gravis grade 2-4;
  8. Guillain-Barre syndrome (GBS) or transverse myelitis of any grade;
  9. Grade 2-4 encephalitis;
  10. Severe or life-threatening grade 3-4 pancreatitis;
  11. Severe or life-threatening bullous disease (grade 3-4);
  12. Severe grade 3-4 uveitis or episcleritis;
* Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation or long-term corticosteroid therapy. Patients with thyroid, suprarenal or hypopituitarism that could be controlled only with hormone replacement therapy, type 1 diabetes mellitus, psoriasis or vitiligo without systemic treatment, etc., were eligible to participate in the study.
* Non-resolution of toxicity after previous antineoplastic therapy, i.e., resolution to baseline, NCI-CTCAE 5.0 grade 0-1 (excluding alopecia), or inclusion/exclusion criteria. Irreversible toxicities (e.g., hearing loss) that would not reasonably be expected to be exacerbated by the study drug can be included in the study;
* Known history of clinically significant liver disease, including active viral hepatitis (hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HbcAb) positive, HBV DNA>10000 copies /mL or >2000 IU/mL; Hepatitis C virus (HCV) antibody positive and HCV RNA positive], or other active hepatitis, clinically significant moderate to severe cirrhosis;
* Patients with uncontrolled third space effusion requiring repeated drainage, such as pleural effusion, ascites, pericardial effusion, etc. (Patients who do not need drainage of effusion or stop drainage for 3 days without significant increase in effusion can be enrolled);
* Receiving a systemic corticosteroid (prednisone > 10mg/ day or equivalent) or other immunosuppressive medication within 14 days before the first study medication;
* Patients with any severe and/or uncontrolled disease, including:

  1. Hypertension that is not well controlled by antihypertensive medication (systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg);
  2. Unstable angina pectoris or myocardial infarction, coronary artery bypass grafting or stent implantation within 6 months before study medication;
  3. Grade I or above myocardial ischemia or myocardial infarction, arrhythmia (including QTc≥480ms) and ≥ grade 2 congestive heart failure (New York Heart Association (NYHA) classification); Degree Ⅱ or above heart block; Left ventricular ejection fraction (LVEF) < 50%;
  4. Poorly controlled diabetes (fasting blood glucose > 10 mmol/L);
  5. Patients with urinary protein ≥++ and confirmed 24-hour urinary protein > 1.0g;
  6. Severe active or uncontrolled infection;
* Patients with or suspected to have active autoimmune diseases, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, etc.;
* Renal failure requiring hemodialysis or peritoneal dialysis;
* Patients with a history of immunodeficiency, including HIV positive patients, other acquired immunodeficiency diseases, congenital immunodeficiency diseases, or organ transplantation history;
* History of live attenuated vaccine inoculation within 4 weeks before the first study drug or the expected vaccination during the study period;
* History of psychiatric drug abuse and can not quit or have a history of mental disorders;
* The presence of any other severe, acute or chronic medical disease or mental illness or laboratory abnormality, as judged by the investigator, that may increase the risk associated with participation in the study or that may interfere with the interpretation of the results of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Immune-related pathologic reponse rate (irPR） | Date of surgery
  IrPR is defined as the proportion of patients achieving a complete pathologic or major pathologic response. Complete or major pathological response are assessed according to the proportion of viable residual tumor in the initial tumor bed of HE sections from tumor tissue. Complete pathological response means no viable residue tumor in the initial tumor bed, and major pathological response with a ≤10% viable residue tumor in the initial tumor bed.

SECONDARY OUTCOMES:
Adverse events | From first dose to 28 days after last dose
  The number of participants experiencing adverse events according to Common Terminology Criteria for Adverse Events version 5.0 (CTCAE 5.0). The safety profile of the treatment will be documented and summarized by summary statistics as frequency and percentage for each AE.
Surgical morbidity | From date of surgery up to 28 days after surgery
  Surgical morbidity is assessed by Clavien-Dindo classification.
Objective response rate (ORR) | Baseline to date of surgery
  Tumor response rate is assessed respectively according to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1). ORR is defined as the proportion of patients who are evaluated as CR and PR.
Imaging density changes of lesions | Baseline to date of surgery
  Patients will undergo baseline and preoperative contrast-enhanced CT scans. In the portal venous phase, the margins of the primary and metastatic lesions will be outlined, and their average CT values will be calculated to reflect the change in density at a time.
Down-staging rate of primary tumor T staging | Baseline to date of surgery
  The T stage of the primary tumor will be evaluated according to the AJCC criteria at baseline and before surgery to reflect the change in T stage of the primary tumor after preoperative treatment.
Rate of distant metastasis | Up to 2 years after surgery. Patients will be followed every 3 months the 1st year, and every 6 months the next year.
  At postoperative follow-up, the number and timing of patients who developed distant metastases will be recorded. This endpoint focuses on patients in cohort 1 and 2.
Progression free survival (PFS) | Up to 2 years after surgery. Patients will be followed every 3 months the 1st year, and every 6 months the next year.
  PFS is defined as the time from the first dose of neoadjuvant theratpy to progression disease or death from any cause, whichever occurs first.

OTHER OUTCOMES:
Peripheral plasma and tissue-based biomarker analysis | Up to 2 years after start of treatment
  Punctured tumor tissue and surgical resection samples were collected for revealing changes in the tumor microenvironment. Baseline, post-treatment, and postoperative plasma for revealing changes in peripheral blood biomarkers.

CONTACTS AND LOCATIONS:
Locations (1):
- Jinling Hospital, Affiliated Hospital of Medical School, Nanjing University, Nanjing, China, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No